CLINICAL TRIAL: NCT04006249
Title: Haemochromatosis and Periodontitis
Acronym: HEMOPARO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-A00998-49
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: to Evaluate the Prevalence of Periodontal Diseases in Patients With Hemochromatosis at the Time of Diagnosis and / or Their Usual Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diagnostic test (Other)
  Interventions: Diagnostic Test: dental probes

INTERVENTIONS:
Diagnostic Test: dental probes — Measurement of the depth of the periodontal pockets and clinical loss

SUMMARY:
Periodontitis is a chronic inflammatory disease that affects tissues surrounding the teeth. It is strongly associated with the major pathogenic "red complex", including Porphyromonas gingivalis, Tannerella forsythia and Treponema denticola1 and thus is considered an infection. Recent advances in the pathogenesis of periodontal disease have suggested that polymicrobial synergy and microbiota dysbiosis together with a dysregulated immune response can induce inflammation-mediated damage in periodontal tissues2-4. Interestingly, currently periodontitis is associated with a growing number of systemic diseases, including cardiovascular diseases, adverse pregnancy outcomes, diabetes5-7 and hereditary haemochromatosis8.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 35 to 64 years with homozygosity hemochromatosis C282Y
* Patients regularly enrolled in a health insurance plan
* Patients with at least 10 natural teeth
* Patients who have given informed written, dated and signed consent

Exclusion Criteria:

* Diabetic patients
* Simultaneous participation in another study
* Pregnant or lactating women
* The incapacitated persons and persons deprived of their liberty
* Patients who do not speak French, both written and spoken
* Patients previously included in this trial
* Patients with heart valves or endovascular equipment (risk of infective endocarditis ...)
* Patients with a history of maxillofacial surgery
* Patients whose oral status is considered incompatible with entry into the study, at the discretion of the investigator
* Patients on drugs that can cause gingival hypertrophy, such as Hydantoins (phenytoin), Dihydropyridines, Diltiazem or Ciclosporin
* Patients on medication that can cause gingival bleeding (anticoagulants, antiplatelet agents and aspirin).

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2010-06-06 (Actual); Primary Completion 2011-09-22 (Actual); Study Completion 2011-12-01 (Actual)

PRIMARY OUTCOMES:
prevalence of periodontal diseases | 2 years
  To evaluate the prevalence of periodontal diseases in patients with hemochromatosis at the time of diagnosis and / or their usual therapeutic